CLINICAL TRIAL: NCT00146679
Title: Psychoeducational Intervention for ICD Patients (PEACE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sandra B. Dunbar, RN, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0430-1999; SR01 NR 5187-03
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure; Ventricular Arrhythmias
Keywords: Heart failure; Ventricular arrhythmias; ICD; Psychoeducational intervention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (UC) (Placebo Comparator): Usual Care provided by providers
  Interventions: Behavioral: Usual Care
- Psychoeducational Telephone CounselingTC (Active Comparator): Education and Counseling for ICD patients provided through Telephone Contact
  Interventions: Behavioral: Psychoeducational Telephone counseling (TC)
- Psychoeducation through Groups (SG) (Active Comparator): Education and Counseling for ICD patients provided in a group setting with other ICD Patients
  Interventions: Behavioral: Psychoeducational Intervention by Group (SG)

INTERVENTIONS:
Behavioral: Psychoeducational Telephone counseling (TC) — Educational and Counseling, symptom management training and cognitive behavioral intervention to teach coping skills provided through telephone sessions
  Other Names: TC
  Arms: Psychoeducational Telephone CounselingTC
Behavioral: Psychoeducational Intervention by Group (SG) — Educational and Counseling, symptom management training and cognitive behavioral intervention to teach coping skills provided in 4 group sessions
  Other Names: SG
  Arms: Psychoeducation through Groups (SG)
Behavioral: Usual Care — Usual Care provided by providers
  Other Names: UC
  Arms: Usual Care (UC)

SUMMARY:
The overall purpose of this study is to test the effects of a nurse managed psychoeducational intervention, consisting of symptom management training (SMT) and cognitive-behavioral intervention (CBI), during the first year after ICD implantation using a 3 group randomized clinical trial.

DETAILED DESCRIPTION:
Symptom distress and persistent physical and psychological changes characterize early and ongoing recovery from ventricular dysrhythmia and treatment with an implantable cardiac defibrillator (ICD). This study will test the effect of a psycho educational intervention on psychological and physical outcomes in the first 12 months after ICD implantation. Primary outcome measures are anxiety, depression, and functional status. The effect of the intervention on variables that mediate adaptation and outcomes (symptoms, illness appraisal, and coping behaviors) will also be examined. Secondary aims will examine subsequent arrhythmia events (ICD delivered therapy) and health resource utilization in relation to the main outcomes. The intervention and study variables are based on stress and coping theory and previous research with ICD patients, which documented negative outcomes of ineffective coping and compelling relationships between increased emotional distress and subsequent arrhythmia events.

A three-group, randomized, clinical trial with a repeated-measures design will be used. ICD patients (n=240) will be randomized to receive either the usual standard of care, symptom management training plus cognitive behavioral intervention delivered in a group format, or symptom management training plus cognitive behavioral intervention delivered by nurse provided telephone counseling. The symptom management-training component will be provided in the acute care setting and will focus on symptoms of pain, sleep disturbances and ICD shocks. The four cognitive behavioral sessions by group or telephone format will begin 6-8 weeks after hospitalization and will focus on illness reappraisal and coping skill training. Thus the intervention is designed to bridge the acute and outpatient continuum of care. A booster intervention will be provided at 4 months after implantation. Timeframes for evaluations are baseline, 1, 3, 6, and 12 months after implantation. This study will test whether a cost-effective, accessible, theoretically based, nurse-managed, psycho educational intervention provides an incremental effect over usual care in improving psychological and physical outcomes in ICD patients. This study will provide data upon which future clinical practice guidelines can be based and will establish priorities for patient care according to which interventions are linked to improved adaptive processes and patient outcomes. Greater understanding of the relationships among psychological and physical outcomes, arrhythmia events, and health resource utilization are important for future studies and evaluation of clinical practice with ICD patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a nonthoracotomy insertion
* Have a primary cardiac etiology of their ventricular arrhythmia (coronary artery disease, cardiomyopathy, valve dysfunction, or combination)
* Be fluent in English
* Live within a 75 mile radius of the coordinating center
* Be accessible by telephone
* Only those receiving their first ICD, not replacement generators, will be entered.

Exclusion Criteria:

* Being evaluated or on a waiting list for heart transplantation
* Congenital disease or long QT syndrome
* Disorientation documented in the pre-implantation hospitalization period
* History of psychiatric disorder or progressively debilitating comorbidity that would confound outcome measures

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2001-03; Primary Completion 2005-06 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Anxiety | 3, 6, 12 months
  State-Trait Anxiety Inventory (STAI)
Depression | 3, 6, 12 months
  Beck Depression Inventory II
Functional status | 3, 6, 12 months
  Duke Activity Status Index

SECONDARY OUTCOMES:
Subsequent arrhythmia events documented by ICD therapy | 3, 6, 12 months
  Arrhythmia events log
Patterns of health resource utilization (re-hospitalization, scheduled and unscheduled outpatient visits and contacts, disability days) | 3, 6, 12 months
  Health Resource Use Questionnaire (HRUQ)
Coping | 3, 6 12 months
  Jalowiec Coping Scale
Symptoms | 3,6, 12 months
  Brief Pain Inventory and Pittsburgh Sleep Quality Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B. Dunbar, RN, DSN, Principal Investigator — Emory University School of Nursing
Locations (5):
- United States (5):
  - Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia

REFERENCES:
- [Background] Dunbar SB. Psychosocial issues of patients with implantable cardioverter defibrillators. Am J Crit Care. 2005 Jul;14(4):294-303. PMID 15980420
- [Background] O'Brien MC, Langberg J, Valderrama AL, Kirkendoll K, Romeiko N, Dunbar SB. Implantable cardioverter defibrillator storm: nursing care issues for patients and families. Crit Care Nurs Clin North Am. 2005 Mar;17(1):9-16, ix. doi: 10.1016/j.ccell.2004.09.002. PMID 15749396
- [Background] Dunbar SB, Funk M, Wood K, Valderrama AL. Ventricular dysrhythmias: nursing approaches to health outcomes. J Cardiovasc Nurs. 2004 Sep-Oct;19(5):316-28. doi: 10.1097/00005082-200409000-00007. PMID 15495892
- [Result] Berg SK, Higgins M, Reilly CM, Langberg JJ, Dunbar SB. Sleep quality and sleepiness in persons with implantable cardioverter defibrillators: outcome from a clinical randomized longitudinal trial. Pacing Clin Electrophysiol. 2012 Apr;35(4):431-43. doi: 10.1111/j.1540-8159.2011.03328.x. Epub 2012 Feb 3. PMID 22303998
- [Result] Dunbar SB, Langberg JJ, Reilly CM, Viswanathan B, McCarty F, Culler SD, O'Brien MC, Weintraub WS. Effect of a psychoeducational intervention on depression, anxiety, and health resource use in implantable cardioverter defibrillator patients. Pacing Clin Electrophysiol. 2009 Oct;32(10):1259-71. doi: 10.1111/j.1540-8159.2009.02495.x. PMID 19796343
- [Result] Smith G, Dunbar SB, Valderrama AL, Viswanathan B. Gender differences in implantable cardioverter-defibrillator patients at the time of insertion. Prog Cardiovasc Nurs. 2006 Spring;21(2):76-82. doi: 10.1111/j.0889-7204.2006.04843.x. PMID 16760689
- See also: LInk to PubMed reference site for Berg, SK et al 2012 — http://www.ncbi.nlm.nih.gov/pubmed/22303998
- See also: link to PubMed reference for study results by Dunbar, SB et al 2009 — http://www.ncbi.nlm.nih.gov/pubmed/19796343